CLINICAL TRIAL: NCT00534378
Title: Phase I, Open-Label, Single-Center Study to Evaluate the Safety and Dose Linearity of Intramuscular Administration of Midazolam Using
Brief Title: Phase I Trail for Intramuscular Administration of Midazolam Using An Autoinjector
Acronym: AAS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Office of the Surgeon General (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11903
Record Dates: First submitted 2007-09-20; First posted 2007-09-24 (Estimated); Last update posted 2007-09-24 (Estimated); Status verified 2007-09

CONDITIONS: Seizures
Keywords: Nerve agent; Midazolam; Seizures; Severe recurrent convulsive seizures induced by nerve agent exposure
MeSH Terms: conditions — Seizures | interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (No Intervention)
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Midazolam — The study drug was administered IM into the anterior thigh using the preloaded autoinjector. The autoinjectors were preloaded with midazolam 5 mg or 10 mg with a total volume of 1 or 2 mL. Healthy subjects were assigned to one of six target dosage groups (0.10, 0.18, 0.25, 0.33, 0.40, 0.49 mg/kg) and, based on their weight, received the necessary combination of fixed 5 or 10 mg doses to provide the assigned target dose.

SUMMARY:
Purpose of the study is to determine midazolam's safety and dose-linearity when delivered intramuscularly via an autoinjector. The proposed initial treatment dosage for seizures induced by exposure to nerve agents.

DETAILED DESCRIPTION:
The investigational drug product being evaluated in this study is the Midazolam Autoinjector. This system is composed of an autoinjector filled with the drug product midazolam EP. The study drug is administered IM into the anterior thigh using the preloaded autoinjector. This method of administration was selected as it is the method that will be used in later clinical trials and for the marketed product. The autoinjectors were preloaded with midazolam 5 mg or 10 mg with a total volume of 1 or 2 mL. Healthy subjects are assigned to one of six target dosage groups (0.10, 0.18, 0.25, 0.33, 0.40, 0.49 mg/kg) and, based on their weight, received the necessary combination of fixed 5 or 10 mg doses to provide the assigned target dose.

ELIGIBILITY:
Inclusion Criteria:

* Generally health adult
* Physically fit
* Body Mass Index of >/- 19 and </- 26 and a body weight of 55 to 85 Kg
* Have adequate venous access and sufficient upper leg muscle tissue
* Have all specified laboratory values
* Have a negative assay for HIV-1, HIV-2, HbsAg
* If femal is of child bearing potential, she must not be pregnant or breast feeding, nor plan to become pregnant for th eduration of the study. She must have a negative blood serum pregnancy test within 21 days of treatment, and a negative urine pregnancy test prior to dosing.
* Females of childbearing potential will use adequate contraception.
* Willing to refrain from donating blood for 8 weeks after compeletion of the study.

Exclusion Criteria:

* Participated in a pharmacokinetic study or any clinical study currently or within the last 30 days or donated >480mL of blood within the last 8 weeks.
* History or presence of significant cardiovascular, hepatic, renal, hematologic, gastrointestingal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease that could potentially impact the safety of the subject or metabolism of the drug.
* Be taking any medications to ttreat a chronic medical condition
* Have ongoing drug abuse/dependence (including alcohol); or history of or treatment for alcohol or drug abuse
* History of allergic or untoward reaction to any benzodiazepine or any psychotropic agent
* Currently suffering frm acute or chronic pulmonary disease
* Clinically relevant abnormal history, physical findings, ECG, or laboratory values at the pre-study screening assessment that could interfere with objectives of the study or the safety of the subject.
* Pregnant or nursing
* History of glaucoma
* Positive urine test for drug abuse
* Have an active malignancy or history of metastatic or hematologic malignancy with the exception of melanoma in situ or basal or squamous cell carcnoma of the skin Subjects with positive tests for hepatitis B, hepatitis C, syphilis, HIV-1 or HIV-2
* Subjects whoe ECG reveals a PR interval >/- 190 msec
* Subjects should refrain from taking any OTC preparations, herbal remedies, and/or nutritional supplement taken within 7 days prior to study drug drug administration.
* Subjects not using medically recognized means of birth control
* Subjects with a prior history of seizures or related conditions

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2006-07; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Holohan, MD, Principal Investigator — Bioanalytical Systems, Inc.
Locations (1):
- BASi Baltimore Clinical Research Unit, Baltimore, Maryland, United States